CLINICAL TRIAL: NCT07010653
Title: Dilapan-S Versus Double Balloon Catheter (CRB) for Preinduction of Labor at Term
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Giuseppe Rizzo, Prof. Giuseppe Rizzo, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 400/8.04.2025 4a3
Record Dates: First submitted 2025-05-12; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Induction of Labor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dilapan-S (Experimental): Dilapan-S Participants assigned to the Dilapan-S group will have 3 to 5 rods inserted under aseptic conditions. Placement will follow manufacturer instructions, and rods will remain in place for up to 12 hours unless spontaneous labor or device expulsion occurs earlier. Upon removal, cervical status will be assessed, and induction will continue with prostaglandins or oxytocin based on standard care
  Interventions: Device: Higroscopic Cervical ripening
- Double Balloon Catheter (CRB) (Active Comparator): Participants randomized to CRB will undergo insertion of a double balloon catheter with inflation of each balloon (approximately 80 mL saline each) according to established protocols. The catheter will remain for up to 12 hours or until spontaneous labor or expulsion. Post-removal management will mirror that of the Dilapan-S group.
  Interventions: Device: Cervical ripening via CRB

INTERVENTIONS:
Device: Higroscopic Cervical ripening — Participants assigned to the Dilapan-S group will have 3 to 5 rods inserted under aseptic conditions. Placement will follow manufacturer instructions, and rods will remain in place for up to 12 hours unless spontaneous labor or device expulsion occurs earlier. Upon removal, cervical status will be assessed, and induction will continue with prostaglandins or oxytocin based on standard care.
  Arms: Dilapan-S
Device: Cervical ripening via CRB — Double Balloon Catheter (CRB) Participants randomized to CRB will undergo insertion of a double balloon catheter with inflation of each balloon (approximately 80 mL saline each) according to established protocols. The catheter will remain for up to 12 hours or until spontaneous labor or expulsion. Post-removal management will mirror that of the Dilapan-S group.
  Arms: Double Balloon Catheter (CRB)

SUMMARY:
Induction of labor (IOL) is a frequently performed procedure in obstetrics, aimed to achieve vaginal delivery when continuing the pregnancy is no longer advisable. A key determinant of IOL success is cervical ripening, particularly when the cervix is initially unfavorable. A range of preinduction methods is available, encompassing both mechanical and pharmacological approaches. Among mechanical techniques, the double balloon catheter (CRB) facilitates cervical dilation by applying direct pressure, which stimulates local prostaglandin release. In contrast, Dilapan-S, a synthetic osmotic dilator, works by gradually expanding through the absorption of cervical fluids, thereby applying gentle mechanical pressure.

While both methods are widely used and generally considered safe, there is limited evidence directly comparing their effectiveness and patient-centered outcomes. Mechanical methods are associated with a lower risk of uterine hyperstimulation compared to pharmacological alternatives. The choice between CRB and Dilapan-S may significantly influence labor duration, cesarean delivery rates, maternal comfort, and hospital resource utilization. This study aims to fill the existing knowledge gap by directly comparing Dilapan-S and CRB for term preinduction, with a focus on clinical efficacy and maternal satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* • Singleton pregnancy

  * Cephalic fetal presentation
  * Gestational age ≥ 37+0 weeks
  * Indication for labor induction (e.g., postdates, maternal hypertension)
  * Bishop score ≤ 6
  * Maternal age ≥18 years
  * Ability to provide informed consent

Exclusion Criteria:

* • Premature rupture of membranes (PROM)

  * Placenta previa, vasa previa, or abnormal placentation
  * Active genital tract infection
  * Prior classical cesarean section or extensive uterine surgery
  * Known fetal anomaly contraindicating vaginal delivery
  * Allergy or sensitivity to device materials
  * Any contraindication to labor induction or vaginal birth

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Time from initiation of cervical ripening to time of delivery measure in hours and minutes | from the time of beginning of cervical ripening to the time of delivery measure in hours and minutes

SECONDARY OUTCOMES:
Change in Bishop score after device removal | From the time of beggining of cervical ripening to the time of removal of the device (CRB or dilapan S) 12 hours
  Bishop score scaled from 0 to 10 (higher values indicated better cervical ripening)
Mode of delivery | at the time of delivery
  spontaneous vaginal delivery, operative vaginal delivery, emergency cesarean delivery
Need for additional ripening agent | From removal of CRB or dilapanS to 96 hours after enrollment
  after the removal of CRB or dilapanS needs of using misoprol or dinoprostone to complete cervical ripening
Maternal discomfort assessed by VAS | from CRB insertion or DilapanS removal (12 hours)
  Pain was assessed using the Visual Analog Scale (VAS), ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst imaginable pain. Higher scores represent worse outcomes.
Apgar Score | at the time of delivery
  0 to 10 (10 better newborn cindition)
NICU admission | From delivery to 28 days of life of the newborn
Chorioamnionitis | From enrollment to 6 weeks postpartum
Uterine Tachysystole | From enrollment to delivery (duration of labor measured in hours)
  number of uterine contractions every 10 minutes measured
Changes in fetal heart rate trace | From enrollment to delivery (labor measured in hours)
  changes in fetal heart baseline, variability, presence of deceleration
Postpartum hemorrhage | From delivery to the first day (hours(
  blood loss > 500 ml for spontaneous delivery; > 1000 ml for cesarean delivery

IPD SHARING:
Plan to Share IPD: Undecided